CLINICAL TRIAL: NCT04624880
Title: COMT Activity as a Biomarker for Hypnotizability and Hypnotic Analgesia Using a Multiplexed Precision Medicine Platform
Brief Title: COMT Activity and Hypnotizability
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jessie Kittle, Assistant Professor of Medicine, Stanford University
Other Study IDs: 58341
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Genetic Predisposition
Keywords: Hypnosis; Biosensing, technique; Pain, psychology; Analgesia,psychology; Hypnotizability; Giant Magnetoresistive Sensors
MeSH Terms: conditions — Pain, Postoperative; Genetic Predisposition to Disease; Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva samples for DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Participants with HIP previously measured: This cohort of patients will have their genetics analyzed and compared to their HIP scores.
  Interventions: Device: Giant magnetoresistive sensor (GMR)
- Participants without HIP measured: This cohort of patients from the control group of the knee replacement trial (who did not have their HIP measured) will have their genetics, pain, and opioid use analyzed, and compared to the genetics, pain, and opioid use of the hypnosis group from that trial.
  Interventions: Device: Giant magnetoresistive sensor (GMR)

INTERVENTIONS:
Device: Giant magnetoresistive sensor (GMR) — Giant magnetoresistive sensor analyzes genetic polymorphisms in patient samples.

SUMMARY:
Hypnosis is an effective pain management tool for surgery that can reduce opioid use up to 40%. COMT single nucleotide polymorphisms (SNPs) can predict pain sensitivity and opioid use perioperatively, and may also be associated with hypnotizability or response to hypnotic analgesia. Analyzing COMT haplotypes from DNA extracted from saliva or blood using a giant magnetoresistive (GMR) nanotechnology platform may be faster, less expensive, and at least as accurate as pyrosequencing. This study aims to validate a multi-SNP point-of-care (POC) GMR assay for the rapid genotyping of SNPs predictive of COMT activity, and test the feasibility of using COMT activity as a biomarker for hypnotizability and/or response to hypnotic analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in one of 3 specific hypnosis trials
* Enrollment is by invitation only

Exclusion Criteria:

* Participants in the prior trials who declined to be contacted for future research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this trial are drawn from three prior trials. One trial measured hypnotizability and collected genetic samples with permission to use for future research, 23 samples will be drawn from this cohort. The second trial measured hypnotizability in healthy volunteers, 42 participants agreed to be contacted for future studies will be invited to participate by submitting a saliva sample for DNA analysis. The third trial used hypnotic analgesia for knee replacement surgery, approximately 32 patients had hypnotizability tested and will be invited to participate for the primary analysis. Another approximately 30 patients from the control group of that trial had pain and opioid use collected postoperatively, and will be invited to provide genetic sample to be used for the secondary outcome analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Percent concordance of rapid genotyping of SNPs with giant magnetoresistive sensors vs. genotyping using pyrosequencing | Through study completion, average of 2 years
  We will test the hypothesis that the four COMT SNPs (rs4680, rs4818, rs4633, and rs6269) can be detected on the GMR platform with 99% accuracy when compared to pyrosequencing
Determine which COMT SNP haplotypes associate with high/medium/low hypnotizability measured by the Hypnotic Induction Profile score. | Through study completion, average of 2 years

SECONDARY OUTCOMES:
Determine which COMT diplotypes/haplotypes associate with high/medium/low postoperative opioid use in milligram morphine equivalents/hour/kilogram of body weight (MME/kg/hr), and high/medium/low average pain scores on the Numeric Pain Scale. | Through study completion, average of 2 years
  Determine if there is a relationship between COMT diplotypes/haplotypes and pain or opioid use in a subgroup of patients who underwent hypnosis prior to knee replacement surgery vs. patients in the control group who were not hypnotized, during their inpatient admission postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Shan Wang, PhD, Principal Investigator — Stanford University; David Spiegel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University/Stanford Healthcare, Palo Alto, California, United States